CLINICAL TRIAL: NCT00675428
Title: A Phase 1/2, Two-Arm, Dose-Finding Study of Natalizumab for the Treatment of Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: Study of Natalizumab in Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision due to low enrollment and not safety concerns.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101MY201
Record Dates: First submitted 2008-05-06; First posted 2008-05-09 (Estimated); Results first posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Multiple Myeloma
Keywords: Relapsed or refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Natalizumab 300 mg (Experimental): Intravenous (IV) infusions of natalizumab 300 mg once every 28 days for 6 months.
  Interventions: Drug: BG00002 (natalizumab)
- Natalizumab 450 mg (Experimental): Intravenous (IV) infusions of natalizumab 450 mg once every 28 days for 6 months.
  Interventions: Drug: BG00002 (natalizumab)

INTERVENTIONS:
Drug: BG00002 (natalizumab)
  Other Names: Tysabri

SUMMARY:
The primary objectives of the study are to evaluate the safety profile and the anti-tumor activity of 2 dose levels of natalizumab in participants with relapsed or refractory multiple myeloma. Secondary objectives are to assess the pharmacokinetic (PK) profile of natalizumab in this study population and to assess peripheral blood mononuclear cell (PBMC) saturation of very late antigen-4 (VLA-4, an α4-integrin) and evaluate possible correlations with clinical activity.

DETAILED DESCRIPTION:
Despite no protocol-defined study stopping criteria being met, the sponsor decided to terminate enrollment after the phase 1 portion was complete and to not move into the phase 2 portion of the study. This decision was made due to difficulty enrolling participants and was not due to any safety concerns.

ELIGIBILITY:
Key Inclusion Criteria:

* Relapsed or refractory multiple myeloma that was treated with or was considered inappropriate for treatment with bortezomib and an IMiD® drug (including an analogue).
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤2.
* Corrected calcium <10.6 mg/dL.

Key Exclusion Criteria:

* Candidates for stem cell transplantation willing to undergo transplantation. (Subjects who are candidates for stem cell transplantation, but are not willing to undergo transplant will be eligible for the study.)
* Autologous stem cell transplantation <3 months post-transplant.
* Prior allogeneic stem cell transplantation.
* Nonsecretory myeloma.
* Plasma cell leukemia (>2000/µL circulating plasma cells by standard cell counting differential), hyperleukocytosis (white blood cells >100,000/µL), clinical evidence of hyperviscosity syndrome, or polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes syndrome (POEMS), or primary systemic amyloidosis.
* Subjects who cannot undergo a brain magnetic resonance imaging (MRI) study.
* Clinically significant (as determined by the Investigator) 12 lead electrocardiogram (ECG) abnormalities, including QTc prolongation (>450 ms in males, >470 ms in females).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (2):
- United States (2):
  - Research Center, Scottsdale, Arizona
  - Research Center, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This record includes data up to and including the last data values collected during long-term follow-up (27 January 2010).
Period: Overall Study
Arm/Group | Natalizumab 300 mg | Natalizumab 450 mg
Started | 3 | 3
Completed | 0 | 0
Not Completed | 3 | 3
Not completed — Disease Progression | 2 | 2
Not completed — No Disease Response After Cycle 6 | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Natalizumab 300 mg | Natalizumab 450 mg | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Median (Full Range); unit: years] | 67.0 [57 to 75] | 68.0 [50 to 75] | 67.5 [50 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs = any ≥grade 3 toxicity related to treatment; treatment delays of ≥7 days due to any toxicity related to treatment, with the exception of hepatic transaminases; or alanine and/or aspartate aminotransferase (ALT and/or AST) >3*upper limit of normal (ULN) with either a total bilirubin >2*ULN or an international normalized ratio (INR) >1.5 related to treatment, or with the appearance of worsening fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, or eosinophilia.
Time Frame: Day 1 up to Day 28
Measure: Number; unit: participants
Arm/Group | Natalizumab 300 mg | Natalizumab 450 mg
Number analyzed (Participants) | 3 | 3
participants | 0 | 0

2. Primary Outcome: Objective Response Rate (ORR)
Description: Response rates were classified according to the International Uniform Response Criteria for Multiple Myeloma (Durie et al, 2006).
Time Frame: Day 1 up to Month 6
Population: ORR was not calculated because the study was terminated early.
Arm/Group | Natalizumab 300 mg | Natalizumab 450 mg
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered medicinal (investigational) product and that does not necessarily have a causal relationship with this product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. See the adverse events section of the record for more details.
Time Frame: Day 1 up to Month 6
Measure: Number; unit: participants
Arm/Group | Natalizumab 300 mg | Natalizumab 450 mg
Number analyzed (Participants) | 3 | 3
participants | 3 | 3

4. Secondary Outcome: Number Of Participants Who Achieve A Complete Response
Description: Response rates were classified according to the International Uniform Response Criteria for Multiple Myeloma (Durie et al, 2006). Complete Response (CR): negative immunofixation on the serum and urine, and disappearance of any soft tissue plasmacytomas , and ≤ 5% plasma cells in the bone marrow. Stringent CR (sCR): CR as defined above, and normal free light chain (FLC) ratio, and absence of clonal cells in the bone marrow by immunohistochemistry or immunofluorescence, based on a κ/λ ratio of > 4:1 or < 1:2 performed on a minimum of 100 plasma cells.
Time Frame: Day 1 up to Month 6
Measure: Number; unit: participants
Arm/Group | Natalizumab 300 mg | Natalizumab 450 mg
Number analyzed (Participants) | 3 | 3
participants | 0 | 0

5. Secondary Outcome: Kaplan-Meier Estimates for Duration Of Response For Participants With A Response
Description: Response rates were classified according to the International Uniform Response Criteria for Multiple Myeloma (Durie et al, 2006). Kaplan-Meier methods were used to estimate the median duration of response and associated 95% confidence intervals.
Time Frame: Day 1 up to Month 6
Population: Duration of response was not calculated because the study was terminated early.
Arm/Group | Natalizumab 300 mg | Natalizumab 450 mg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Pharmacokinetic (PK) Profile Of Natalizumab
Description: PK modeling, either compartmental or noncompartmental-based, was used to describe serum concentrations. Standard PK parameters estimated include: area-under-the-concentration-time curve (AUC), maximum-observed concentration (Cmax), time-to-reach maximum concentration (Tmax), total body clearance (Cl), volume of distribution (Vd), and elimination half-life (t1/2).
Time Frame: Cycles 1 and 6: Day 1 (before infusion and 0.25, 2, 6 and 24 hours after infusion), Days 8, 15, 22. Cycles 2-5: Day 1 (before infusion and 0.25 hour after infusion)
Population: PK analysis was not performed because the study was terminated early.
Arm/Group | Natalizumab 300 mg | Natalizumab 450 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Natalizumab Binding Saturation Of α4 Integrin Sites On Peripheral Blood Mononuclear Cells (PBMC)
Time Frame: Cycle 1: Day 1 (1 hour before infusion and 1 and 24 hours after infusion), Days 8, 15, 22. Cycles 2-5: 1 hour before and 1 hour after infusion). Cycle 6: Day 1 (1 hour before infusion and 1 hour after infusion), Days 8, 15, 22.
Population: Analysis of binding saturation of α4 integrin sites was not performed because the study was terminated early.
Arm/Group | Natalizumab 300 mg | Natalizumab 450 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 463 days (from date of first treatment on 4 September 2008 until the Last Patient Last Visit on 10 December 2009).
Arm/Group | Natalizumab 300 mg | Natalizumab 450 mg
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab 300 mg (N=3) | Natalizumab 450 mg (N=3)
Pneumonia (Infections and infestations) | 1 | 0
Acute Renal Failure (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Natalizumab 300 mg (N=3) | Natalizumab 450 mg (N=3)
Pneumonia (Infections and infestations) | 1 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.